CLINICAL TRIAL: NCT00715546
Title: Phase 1 Study of Autologous-Derived Stem Cell Transplantation in Patients With Lipodystrophy
Brief Title: Autologous Adipose-Derived Stem Cell Transplantation in Patients With Lipodystrophy
Acronym: AADSCTPL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Eduardo Mainieri Chem, Phd, Irmandade Santa Casa de Misericórdia de Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISCMPA 1642/07
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2009-03

CONDITIONS: Lipodystrophy
Keywords: Adipose-derived stem cell; Lipodystrophy
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: autologous transplantation of liposuction material enriched with adipose-derived stem cells — Lipoinjection enriched with adipose-derived stem-cells.

SUMMARY:
The aim of this study is to determine the safety of the autologous transplantation of adipose-derived stem cells in the treatment of lipodystrophies.

ELIGIBILITY:
Inclusion Criteria:

* lipodystrophies with necessity of fat grafting
* accept to participate of the study

Exclusion Criteria:

* HIV infection
* Metastatic malignancy
* Body mass index < 20 kg/m²
* Other severe systemic disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2011-08 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of the transplanted area. | one year

SECONDARY OUTCOMES:
Presence of neovascularization, adipose transplantation reabsorption, tissue viability | one year

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo M. Chem, MD, Principal Investigator — Irmandade Santa Casa de Misericórdia de Porto Alegre
Locations (1):
- Irmandade Santa Casa de Misericórdia, Porto Alegre, Rio Grande do Sul, Brazil